CLINICAL TRIAL: NCT01896674
Title: Value of Knowledge-based Iterative Model Reconstruction at Low-kilovoltage Cardiac 256-slice CT: A Comparison of Filtered Back Projection-, Hybrid-, and Iterative Model Reconstruction
Brief Title: Knowledge-based Iterative Model Reconstruction at Low-kilovoltage (kV) Cardiac Computed Tomography (CT)
Status: Completed | Type: Observational
Sponsor: Kumamoto University (Other)
Responsible Party: Principal Investigator, Daisuke Utsunomiya, Lecturer, Kumamoto University
Other Study IDs: Kuma1478
Record Dates: First submitted 2013-07-08; First posted 2013-07-11 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-07

CONDITIONS: Coronary Artery Disease
Keywords: Computed tomography
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study was to compare FBP-, hybrid IR-, and IMR techniques to assess their role in the identification of coronary artery disease and abnormalities in cardiac structures.

ELIGIBILITY:
Inclusion Criteria:

* A BMI of 27 kg/m2 or less and a coronary calcium score of less than 1,000 Agatston units.

Exclusion Criteria:

* BMI exceeded 27 kg/m2
* renal dysfunction (serum creatinine level > 1.5 mg/dl)
* atrial fibrillation
* prior coronary artery bypass grafting
* heart failure (New York Heart Association class III-IV)

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We enroll consecutive patients.
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2012-05; Primary Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Contrast to noise ratio of coronary arteries | 6 months

REFERENCES:
- [Derived] Yuki H, Utsunomiya D, Funama Y, Tokuyasu S, Namimoto T, Hirai T, Itatani R, Katahira K, Oshima S, Yamashita Y. Value of knowledge-based iterative model reconstruction in low-kV 256-slice coronary CT angiography. J Cardiovasc Comput Tomogr. 2014 Mar-Apr;8(2):115-23. doi: 10.1016/j.jcct.2013.12.010. Epub 2014 Jan 12. PMID 24661824